CLINICAL TRIAL: NCT04088084
Title: Effect of Palmitoylethanolamide on Inner Retinal Function in Stable Glaucoma Patients. A Prospective, Randomized, Single Blind, Crossover Clinical Trial by Pattern Electroretinogram.
Brief Title: Effects of Palmitoylethanolamide on Inner Retinal Function in Glaucoma Patients by Pattern Electroretinogram
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Rossi, Gemma Caterina Maria, principal investigator, clinical ophthalmologist, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PEA2015
Record Dates: First submitted 2019-09-06; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — palmidrol

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, prospective, single blind, two treatment and two period crossover study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: examiners were blinded to the assumption or not of PEA in addition to topical therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care+palmitoylethanolamide (Experimental): PEA was supplemented for 3 months to the standard of care (SOC, topical IOP lowering med)
  Interventions: Dietary Supplement: palmitoylethanolamide (PEA) 600 mg
- standard of care (No Intervention): patients were only on topical IOP lowering therapy (SOC)

INTERVENTIONS:
Dietary Supplement: palmitoylethanolamide (PEA) 600 mg — PEA 600 mg was added to topical therapy
  Arms: standard of care+palmitoylethanolamide

SUMMARY:
The general purpose of the study is to evaluate the potential beneficial effects of PEA 600 mg supplementation on RGCs function in subjects with glaucoma by pattern electroretinogram after three months of therapy.

Secondary objectives are to assess effects on intraocular pressure (IOP) values, if any; to record visual acuity, visual field, central corneal thickness (CCT), and Optical coherence tomography (OCT) (ganglion cell complex - GCC) changes, if any and to follow quality of life (QL) perception (general vision -GV and general health - GH of national eye instutute visual functioning questionnaire 25 items - NEI VFQ25)

DETAILED DESCRIPTION:
Monocentric, randomized, prospective, single blind, two treatment and two period crossover study.

The investigators have proposed a cross-over trial to avoid or to detect the bias due to intra-individual variability and because, from preliminary observation, it has been noted that the effects of PEA on pattern-electroretinogram (PERG) are completely reversible after withdrawal, within one month.

The investigators didn't considered a placebo treated group because the patient cannot interfere with the pattern-electroretinogram PERG measurement that is objective and totally patient-independent.

Study duration 12 months Enrolment period 6 months Minimum Follow-up 6 months Start: January, 2015; end January, 2016 Total sample size: 40 patients

ELIGIBILITY:
Inclusion Criteria:

* -age 18 years or older
* diagnosis of primary open angle glaucoma (POAG)
* controlled IOP (<18 mmHg, morning value) with any topical lowering medication (beta-blockers, carbonic anhidrase inhibitors, alpha2agonists, prostaglandin analogues as monotherapy or as associative therapy; betablocker/carbonic anhydrase inhibitor, betablocker/alpha2agonist, prostaglandine/betablocker and alpha2agonist/carbonic anhidrase inhibitor fixed combinations as monotherapy or in association);
* stable IOP<18 mmHg in the last 2 years
* stable disease in the last 2 years (no more than -1 deciBell-dB/year at MD of visual field)
* at least two reliable visual fields per year in the last 2 years
* no filtering surgery or other ocular surgery in the preceding 6 months
* written consent to participate to study procedures and data utilization in an anonymous form

Exclusion Criteria:

* ocular hypertension with normal optic nerve and visual field
* contraindication to PEA
* glaucomatous scotomas within 10 degree from fixation
* any condition limiting the patient's ability to participate in the study;
* other causes of visual field changes, such as cataract, myopic chorioretinopathy, macular diseases, retinal vascular occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
To assess effects of PEA 600 mg a tablet a day on pattern electroretinogram PERG examination at three months of therapy. | 3 months
  changes in amplitude (microVolt) and changes in latency (millisecond) of p50 and n95 waves

SECONDARY OUTCOMES:
To assess effects of PEA 600 mg on intraocular pressure (IOP) values | 3 months
  IOP measure in mmHg
To record visual field changes | 3 months
  changes in MD (deciBell-dB) and pattern standard deviation-PSD (deciBell-dB) of visual field parameters
To follow quality of life - QL - perception using the 25 item National Eye Institute - Visual Functioning Questionnaire (NEI VFQ25) | 3 months
  changes in the total mean score, in the General vision -GV- and in the general health -GH- subscales scores (scores are presented as a number, higher numbers reflect higher QL)

CONTACTS AND LOCATIONS:
Overall Officials: gemma caterina maria rossi, md, Principal Investigator — clinica oculistica

IPD SHARING:
Plan to Share IPD: Yes
data will be published on peer review journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: upon publication
Access Criteria: actually not available

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT04088084/Prot_SAP_000.pdf